CLINICAL TRIAL: NCT04894903
Title: Effects of a Patient Portal Intervention to Address Diabetes Care Gaps: A Pragmatic Randomized Controlled Trial
Brief Title: Effects of a Patient Portal Intervention to Address Diabetes Care Gaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 212257; R18DK123373 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Self-efficacy; Patient Web Portals; Health Information Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients have access to an existing patient web portal (My Health at Vanderbilt) embedded with the Diabetes Care Gaps Patient Portal Intervention.
  .
  Interventions: Other: Diabetes Care Gaps Patient Portal Intervention
- Usual Care (No Intervention): Patients will have access to an existing patient web portal (My Health at Vanderbilt) NOT embedded with the intervention (i.e., usual care).

INTERVENTIONS:
Other: Diabetes Care Gaps Patient Portal Intervention — The Diabetes Care Gaps Patient Portal Intervention is embedded within an existing patient web portal (My Health at Vanderbilt). The intervention (a) notifies patients when selected, clinically meaningful, evidence-based diabetes monitoring & preventative care (e.g., annual urine microalbumin) are due and (b) allows patients to initiate orders for the care.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the effect of a novel patient portal intervention on the number of patients with diabetes care gaps (e.g., no diabetes eye exam i the last 12 months). The intervention is designed to: (a) notify patients when selected, clinically meaningful, evidence-based diabetes monitoring & preventative care (e.g., annual urine microalbumin) are due and (b) allow patients to initiate orders for the care.

DETAILED DESCRIPTION:
Participants will be recruited from 14 VUMC-affiliate adult primary care clinics located throughout Middle Tennessee. Patients will be randomized 1:1 to the intervention or usual care. 500 adult patients with type 1 or 2 diabetes mellitus will be assigned to one of two arms. 250 will be assigned to receive access to the intervention embedded within an existing patient web portal (My Health at Vanderbilt) at Vanderbilt University Medical Center. 250 will be assigned to a usual care comparison arm with access to the currently available version of My Health at Vanderbilt without the study intervention. At enrollment, participants will complete a baseline questionnaire and diabetes health data will be abstracted from the patients' electronic health record (EHR) before being assigned to the intervention or control arm. Participants will receive additional follow-up questionnaires and diabetes health data will be abstracted from the EHR at 3-month, 6-month, and 12-month follow-ups to assess outcomes. In addition, system usage data (user analytics) will be collected throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Established patient with a participating primary care physician from a participating clinic
* Type 1 or 2 diabetes mellitus
* Able to read in English
* Age 18 to 75 years old
* Mobile device (smartphone or tablet) with internet access
* Active My Health at Vanderbilt (MHAV) account

Exclusion Criteria:

* A medical condition that prevents use of a mobile device
* Pregnant or planning to become pregnant during the study period
* Severe difficulty seeing
* On dialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published in a peer-reviewed journal, de-identified individual participant data that underlie the results reported will be available upon requests made to the principal investigator and ending after 36 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data that underlie the results reported will be available after publication in a peer reviewed journal and posted on clinical trials and ending after 36 months after publication.
Access Criteria: Researchers should provide a methodologically sound proposal to achieve their proposed aims. Proposals may be submitted to the principal investigator up to 36 months following publication. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hackstadt AJ, Elasy TA, Gangaputra S, Harper KJ, Mayberry LS, Nelson LA, Peterson NB, Rosenbloom ST, Yu Z, Martinez W. Effects of a Patient Portal Intervention to Address Diabetes Care Gaps: Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2024 Jun 28;13:e56123. doi: 10.2196/56123. PMID 38941148

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 440 patients were enrolled and sent the baseline survey. 433 patients completed the baseline survey. Completion of the baseline survey was required prior randomization and assignment to a study arm.
Groups:
- Intervention: Patients have access to an existing patient web portal (My Health at Vanderbilt) embedded with the Diabetes Care Gaps Patient Portal Intervention.
  Diabetes Care Gaps Patient Portal Intervention: The Diabetes Care Gaps Patient Portal Intervention is embedded within an existing patient web portal (My Health at Vanderbilt). The intervention (a) notifies patients when selected, clinically meaningful, evidence-based diabetes preventative care (e.g., annual urine microalbumin) are due and (b) allows patients to initiate orders for the care.
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 217 | 216
Completed | 213 | 212
Not Completed | 4 | 4
Not completed — Death | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — moved or exited health system | 1 | 3

BASELINE CHARACTERISTICS:
Population: Two participants in the control group were excluded from analysis because they dropped out from the study prior to 3-month data collection. The mixed effects regression analysis requires at least one measurement in the follow-up period. Two individuals dropped out prior the any follow-up data collection and therefore are not included in the study analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 215 | 216 | 431
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 146 | 139 | 285
  >=65 years | 69 | 77 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (12.3) | 58.3 (12.5) | 57.6 (12.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 122 | 107 | 229
  Sex/Gender: Male | 91 | 109 | 200
  Sex/Gender: Other | 1 | 0 | 1
  Sex/Gender: Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 206 | 202 | 408
  Unknown or Not Reported | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 56 | 50 | 106
  Race: White or Caucasian | 143 | 154 | 297
  Race: American Indian or Alaska Native | 1 | 3 | 4
  Race: Asian | 8 | 2 | 10
  Race: Other | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 215 | 216 | 431
eHealth Literacy [Mean (Standard Deviation); unit: units on a scale] — The eHealth Literacy Scale (eHEALS) was used to assess eHealth literacy. The eHEALS is an 8-item survey that uses a 5-point Likert scale, where 1 is "strongly disagree" and 5 is "strongly agree". The eHEALS is scored on a scale of 8-40, with higher scores indicating greater eHealth literacy.
  units on a scale | 33.3 (5.4) | 33.0 (6.0) | 33.1 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diabetes Care Gaps at Baseline, 3 Months, 6 Months, and 12 Months
Description: Number of diabetes care gaps per patient out of four possible:
  1. no diabetes eye exam in the last 12 months,
  2. no hemoglobin A1C blood test in the last 6 months,
  3. no urine microalbumin in the last 12 months, and
  4. no pneumococcal vaccination of any kind ( i.e., never received PPSV-23, PCV-13, PCV-15, or PCV-20) The presence of a diabetes care gap will be assessed by electronic health record (EHR) abstraction.
Time Frame: Baseline, 3-month follow-up, 6-month follow-up, and 12-month follow-up
Population: Two participants in the control group were excluded from analysis because they dropped out from the study prior to 3-month data collection. The mixed effects regression analysis requires at least one measurement in the follow-up period. Two individuals dropped out prior the any follow-up data collection and therefore are not included in the mixed effects regression analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
Participants
  Baseline: No Care Gaps | 75 | 57
  Baseline: One Care Gap | 77 | 79
  Baseline: Two Care Gaps | 37 | 56
  Baseline: Three Care Gaps | 25 | 18
  Baseline: Four Care Gaps | 1 | 6
  3-months follow-up: No Care Gaps | 83 | 91
  3-months follow-up: One Care Gap | 75 | 87
  3-months follow-up: Two Care Gaps | 33 | 26
  3-months follow-up: Three Care Gaps | 18 | 10
  3-months follow-up: Four Care Gaps | 6 | 2
  6-months follow-up: No Care Gaps | 95 | 102
  6-months follow-up: One Care Gap | 71 | 78
  6-months follow-up: Two Care Gaps | 26 | 22
  6-months follow-up: Three Care Gaps | 16 | 12
  6-months follow-up: Four Care Gaps | 7 | 2
  12-months follow-up: No Care Gaps | 89 | 102
  12-months follow-up: One Care Gap | 68 | 69
  12-months follow-up: Two Care Gaps | 36 | 29
  12-months follow-up: Three Care Gaps | 17 | 11
  12-months follow-up: Four Care Gaps | 5 | 5
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p < 0.001, Mixed Models Analysis — This is the calculated p-value. We used an alpha level of 0.05; Adjusted for baseline number of gaps; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.30 to 0.68]

2. Secondary Outcome: Patient Initiated Orders
Description: The number of patient-initiated orders via the study intervention for evidence-based diabetes monitoring and preventative services (e.g., A1c).
Time Frame: 12-month follow-up
Population: This analysis is limited to the intervention arm only because only patients in the intervention arm were able to initiate orders via the study intervention.
Measure: Number; unit: orders initiated
Arm/Group | Intervention
Number analyzed (Participants) | 216
orders initiated
  Hemoglobin a1c | 97
  Urine microalbumin | 107
  Pneumococcal vaccine | 19
  Diabetes eye exam | 46

3. Secondary Outcome: Change in Understanding of Diabetes Monitoring and Preventative Care
Description: Unique study specific items (four items) to assess participant's understanding of measures of diabetes monitoring and preventative care (e.g., Diabetes Eye Exams) will be administered to all study participants. Each multiple-choice item has only one correct answer and the overall measure is scored as the percent of the items answered correctly.
Time Frame: Baseline to 3-month follow-up, baseline to 6-month follow-up, and baseline to 12-month follow-up
Population: Number analyzed varies because not all participants answered all items at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
Participants
  Baseline to 3-months: Recommended frequency of hemoglobin A1C testing: number analyzed (Participants) | 205 | 209
  Baseline to 3-months: Recommended frequency of hemoglobin A1C testing: Correct to Wrong | 13 | 21
  Baseline to 3-months: Recommended frequency of hemoglobin A1C testing: No Change | 170 | 173
  Baseline to 3-months: Recommended frequency of hemoglobin A1C testing: Wrong to Correct | 22 | 15
  Baseline to 6-months: Recommended frequency of hemoglobin A1C testing: number analyzed (Participants) | 209 | 205
  Baseline to 6-months: Recommended frequency of hemoglobin A1C testing: Correct to Wrong | 11 | 16
  Baseline to 6-months: Recommended frequency of hemoglobin A1C testing: No Change | 173 | 171
  Baseline to 6-months: Recommended frequency of hemoglobin A1C testing: Wrong to Correct | 25 | 18
  Baseline to 12-months: Recommended frequency of hemoglobin A1C testing: number analyzed (Participants) | 203 | 200
  Baseline to 12-months: Recommended frequency of hemoglobin A1C testing: Correct to Wrong | 8 | 16
  Baseline to 12-months: Recommended frequency of hemoglobin A1C testing: No Change | 173 | 168
  Baseline to 12-months: Recommended frequency of hemoglobin A1C testing: Wrong to Correct | 22 | 16
  Baseline to 3-months: Recommended frequency of urine microalbumin testing: number analyzed (Participants) | 205 | 209
  Baseline to 3-months: Recommended frequency of urine microalbumin testing: Correct to Wrong | 36 | 37
  Baseline to 3-months: Recommended frequency of urine microalbumin testing: No Change | 141 | 140
  Baseline to 3-months: Recommended frequency of urine microalbumin testing: Wrong to Correct | 28 | 32
  Baseline to 6-months: Recommended frequency of urine microalbumin testing: number analyzed (Participants) | 208 | 202
  Baseline to 6-months: Recommended frequency of urine microalbumin testing: Correct to Wrong | 34 | 28
  Baseline to 6-months: Recommended frequency of urine microalbumin testing: No Change | 144 | 135
  Baseline to 6-months: Recommended frequency of urine microalbumin testing: Wrong to Correct | 30 | 39
  Baseline to 12-months: Recommended frequency of urine microalbumin testing: number analyzed (Participants) | 202 | 199
  Baseline to 12-months: Recommended frequency of urine microalbumin testing: Correct to Wrong | 26 | 32
  Baseline to 12-months: Recommended frequency of urine microalbumin testing: No Change | 142 | 125
  Baseline to 12-months: Recommended frequency of urine microalbumin testing: Wrong to Correct | 34 | 42
  Baseline to 3-months: Recommended frequency of pneumococcal vaccination: number analyzed (Participants) | 204 | 207
  Baseline to 3-months: Recommended frequency of pneumococcal vaccination: Correct to Wrong | 19 | 28
  Baseline to 3-months: Recommended frequency of pneumococcal vaccination: No Change | 149 | 158
  Baseline to 3-months: Recommended frequency of pneumococcal vaccination: Wrong to Correct | 36 | 21
  Baseline to 6-months: Recommended frequency of pneumococcal vaccination: number analyzed (Participants) | 205 | 204
  Baseline to 6-months: Recommended frequency of pneumococcal vaccination: Correct to Wrong | 20 | 27
  Baseline to 6-months: Recommended frequency of pneumococcal vaccination: No Change | 166 | 152
  Baseline to 6-months: Recommended frequency of pneumococcal vaccination: Wrong to Correct | 19 | 25
  Baseline to 12-months: Recommended frequency of pneumococcal vaccination: number analyzed (Participants) | 203 | 198
  Baseline to 12-months: Recommended frequency of pneumococcal vaccination: Correct to Wrong | 19 | 27
  Baseline to 12-months: Recommended frequency of pneumococcal vaccination: No Change | 157 | 151
  Baseline to 12-months: Recommended frequency of pneumococcal vaccination: Wrong to Correct | 27 | 20
  Baseline to 3-months: Recommended frequency of diabetes eye exam: number analyzed (Participants) | 205 | 208
  Baseline to 3-months: Recommended frequency of diabetes eye exam: Correct to Wrong | 6 | 2
  Baseline to 3-months: Recommended frequency of diabetes eye exam: No Change | 193 | 203
  Baseline to 3-months: Recommended frequency of diabetes eye exam: Wrong to Correct | 6 | 3
  Baseline to 6-months: Recommended frequency of diabetes eye exam: number analyzed (Participants) | 208 | 205
  Baseline to 6-months: Recommended frequency of diabetes eye exam: Correct to Wrong | 4 | 2
  Baseline to 6-months: Recommended frequency of diabetes eye exam: No Change | 199 | 200
  Baseline to 6-months: Recommended frequency of diabetes eye exam: Wrong to Correct | 5 | 3
  Baseline to 12-months: Recommended frequency of diabetes eye exam: number analyzed (Participants) | 203 | 200
  Baseline to 12-months: Recommended frequency of diabetes eye exam: Correct to Wrong | 3 | 5
  Baseline to 12-months: Recommended frequency of diabetes eye exam: No Change | 194 | 190
  Baseline to 12-months: Recommended frequency of diabetes eye exam: Wrong to Correct | 6 | 5
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p = 0.29, Mixed Models Analysis; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.20 to 1.62]

4. Secondary Outcome: Change in Confidence Toward Managing Diabetes in General
Description: The 5-item Manage Disease in General Scale of the Chronic Disease Self-Efficacy Scales is a validated measure of the confidence a person has in managing their own health and health care and is closely related to patient activation. The items were adapted to be specific to diabetes rather than a generic condition or illness. Each item uses a 10-point Likert-type scale of response options ranging from 1 (not at all confident) to 10 (totally confident). Responses result in total raw scores ranging from 1 to 10. The score for the scale is the mean of the items. Higher scores indicate greater confidence in managing diabetes in general.
Time Frame: Baseline to 3-month follow-up, baseline to 6-month follow-up, and baseline to 12-month follow-up
Population: Number analyzed varies because not all participants answered all items at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
score on a scale
  Baseline | 8.0 (1.6) | 8.1 (1.5)
  3-month follow-up: number analyzed (Participants) | 203 | 205
  3-month follow-up | 7.9 (1.7) | 7.9 (1.6)
  6-month follow-up: number analyzed (Participants) | 208 | 205
  6-month follow-up | 7.9 (1.7) | 7.9 (1.5)
  12-month follow-up: number analyzed (Participants) | 200 | 198
  12-month follow-up | 7.9 (1.8) | 8.1 (1.7)
  Change baseline to 3-month follow-up: number analyzed (Participants) | 203 | 205
  Change baseline to 3-month follow-up | -0.1 (1.5) | -0.2 (1.4)
  Change baseline to 6-month follow-up: number analyzed (Participants) | 208 | 205
  Change baseline to 6-month follow-up | -0.1 (1.4) | -0.2 (1.3)
  Change baseline to 12-month follow-up: number analyzed (Participants) | 200 | 198
  Change baseline to 12-month follow-up | -0.1 (1.7) | -0.1 (1.3)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p = 0.74, Mixed Models Analysis; beta coefficient = -0.04, 95% CI 2-sided [-0.24 to 0.17]

5. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. The PAID-5 contains 5 items which have a five-point response option (0-4 representing 'Not a problem' through to 'Serious problem'). Total scores on the PAID-5 can range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress care (e.g., Diabetes Eye Exams) will be administered to all study participants.
Time Frame: Baseline to 3-month follow-up, baseline to 6-month follow-up, and baseline to 12-month follow-up
Population: Number analyzed varies because not all participants answered all items at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
score on a scale
  Baseline: number analyzed (Participants) | 214 | 216
  Baseline | 5.5 (4.8) | 5.5 (4.6)
  3-month follow-up: number analyzed (Participants) | 203 | 208
  3-month follow-up | 6.0 (5.1) | 5.8 (5.0)
  6-month follow-up: number analyzed (Participants) | 208 | 203
  6-month follow-up | 5.7 (5.0) | 5.8 (4.8)
  12-month follow-up: number analyzed (Participants) | 203 | 197
  12-month follow-up | 5.1 (4.5) | 5.3 (4.7)
  Change baseline to 3-month follow-up: number analyzed (Participants) | 202 | 208
  Change baseline to 3-month follow-up | 0.4 (3.7) | 0.1 (3.7)
  Change baseline to 6-month follow-up: number analyzed (Participants) | 207 | 203
  Change baseline to 6-month follow-up | 0.2 (3.7) | 0.2 (3.9)
  Change baseline to 12-month follow-up: number analyzed (Participants) | 202 | 197
  Change baseline to 12-month follow-up | -0.2 (3.8) | -0.2 (4.1)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p = 0.88, Mixed Models Analysis; beta coefficient = -0.04, 95% CI 2-sided [-0.60 to 0.51]

6. Secondary Outcome: Satisfaction/Usability of My Health at Vanderbilt
Description: The System Usability Scale (SUS) is a valid measure of usability and assesses user's perceptions of ease of use, likability of the interface, and overall satisfaction. Each question on the 10-item questionnaire is scored on a 5-point Likert scale [0 (Strongly disagree) to 4 (strongly agree)] and the sum is totaled (0-40). The total sum is then multiplied by 2.5 to convert the original scores to a range of 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 85 or above suggests excellent usability. The SUS has been used in several studies of patient facing health information technology (the article describing its psychometric properties has been cited over 500 times) and has excellent internal consistency reliability (Cronbach's alpha of 0.91).
Time Frame: Baseline, 3-month follow-up, 6-month follow-up, and 12-month follow-up
Population: Number analyzed varies because not all participants answered all items at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
score on a scale
  Baseline: number analyzed (Participants) | 210 | 210
  Baseline | 81.3 (13.4) | 80.2 (12.8)
  3-month follow-up: number analyzed (Participants) | 202 | 204
  3-month follow-up | 81.1 (14.3) | 79.4 (14.8)
  6-month follow-up: number analyzed (Participants) | 207 | 203
  6-month follow-up | 82.0 (13.1) | 79.0 (14.8)
  12-month follow-up: number analyzed (Participants) | 200 | 194
  12-month follow-up | 81.6 (14.7) | 80.5 (16.1)
  Change baseline to 3-month follow-up: number analyzed (Participants) | 198 | 198
  Change baseline to 3-month follow-up | -0.1 (14.4) | -0.7 (12.4)
  Change baseline to 6-month follow-up: number analyzed (Participants) | 203 | 197
  Change baseline to 6-month follow-up | 0.6 (12.8) | -1.2 (11.6)
  Change baseline to 12-month follow-up: number analyzed (Participants) | 197 | 188
  Change baseline to 12-month follow-up | 0.3 (13.2) | 0.2 (15.9)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p = 0.21, Mixed Models Analysis; beta coefficient = -1.24, 95% CI 2-sided [-3.19 to 0.71]

7. Secondary Outcome: Change in Blood Glucose Control
Description: Participants' most recent hemoglobin A1C will be abstracted from participants' electronic medical record.
Time Frame: Baseline to 12-month follow-up
Population: Number analyzed differs because not all patients had a qualifying A1c value in the EHR for the timepoint.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
percentage of glycated hemoglobin
  Baseline: number analyzed (Participants) | 212 | 214
  Baseline | 7.0 (1.3) | 7.2 (1.5)
  12-month follow-up: number analyzed (Participants) | 214 | 214
  12-month follow-up | 6.8 (1.4) | 6.9 (1.3)
  Change in Hemoglobin A1C: Baseline to 12-month follow-up: number analyzed (Participants) | 212 | 214
  Change in Hemoglobin A1C: Baseline to 12-month follow-up | -0.17 (1.21) | -0.35 (1.30)

8. Secondary Outcome: Treatment Intensification
Description: The addition of: (a) antihyperglycemic medications and (b) antihypertensive medications will be assessed by EHR abstraction.
Time Frame: Baseline to 3-month follow-up, baseline to 6-month follow-up, and baseline to 12-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
Participants
  Antihyperglycemic medications: baseline to 3-month follow-up: No change in the number of medications | 145 | 163
  Antihyperglycemic medications: baseline to 3-month follow-up: Decrease in the number of medications | 34 | 29
  Antihyperglycemic medications: baseline to 3-month follow-up: Increase in the number of medications | 35 | 24
  Antihyperglycemic medications: baseline to 3-month follow-up: Unknown | 1 | 0
  Antihyperglycemic medications: baseline to 6-month follow-up: No change in the number of medications | 122 | 143
  Antihyperglycemic medications: baseline to 6-month follow-up: Decrease in the number of medications | 47 | 36
  Antihyperglycemic medications: baseline to 6-month follow-up: Increase in the number of medications | 45 | 37
  Antihyperglycemic medications: baseline to 6-month follow-up: Unknown | 1 | 0
  Antihyperglycemic medications: baseline to 12-month follow-up: No change in the number of medications | 103 | 118
  Antihyperglycemic medications: baseline to 12-month follow-up: Decrease in the number of medications | 59 | 51
  Antihyperglycemic medications: baseline to 12-month follow-up: Increase in the number of medications | 52 | 47
  Antihyperglycemic medications: baseline to 12-month follow-up: Unknown | 1 | 0
  Antihypertensive medications: baseline to 3-month follow-up: No change in the number of medications | 190 | 196
  Antihypertensive medications: baseline to 3-month follow-up: Decrease in the number of medications | 11 | 14
  Antihypertensive medications: baseline to 3-month follow-up: Increase in the number of medications | 13 | 6
  Antihypertensive medications: baseline to 3-month follow-up: Unknown | 1 | 0
  Antihypertensive medications: baseline to 6-month follow-up: No change in the number of medications | 184 | 189
  Antihypertensive medications: baseline to 6-month follow-up: Decrease in the number of medications | 15 | 18
  Antihypertensive medications: baseline to 6-month follow-up: Increase in the number of medications | 15 | 9
  Antihypertensive medications: baseline to 6-month follow-up: Unknown | 1 | 0
  Antihypertensive medications: baseline to 12-month follow-up: No change in the number of medications | 162 | 171
  Antihypertensive medications: baseline to 12-month follow-up: Decrease in the number of medications | 26 | 26
  Antihypertensive medications: baseline to 12-month follow-up: Increase in the number of medications | 26 | 19
  Antihypertensive medications: baseline to 12-month follow-up: Unknown | 1 | 0

9. Secondary Outcome: Change in Diabetes Self-efficacy
Description: The Perceived Diabetes Self-Management Scale (PDSMS) is a valid measure of diabetes self-efficacy (i.e., how confident they feel about their ability to carry out multiple self management tasks). The uni-dimensional, 8-item scale is scored on a five-point Likert scale. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Time Frame: Baseline to 3-month follow-up, baseline to 6-month follow-up, and baseline to 12-month follow-up
Population: Number analyzed varies because not all participants answered all items at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 215 | 216
score on a scale
  Baseline: number analyzed (Participants) | 213 | 215
  Baseline | 29.7 (5.6) | 29.8 (5.4)
  3-month follow-up: number analyzed (Participants) | 202 | 206
  3-month follow-up | 29.6 (6.1) | 30.2 (6.2)
  6-month follow-up: number analyzed (Participants) | 207 | 203
  6-month follow-up | 30.0 (6.2) | 30.7 (5.6)
  12-month follow-up: number analyzed (Participants) | 201 | 198
  12-month follow-up | 30.5 (6.2) | 30.8 (6.0)
  Change baseline to 3-month follow-up: number analyzed (Participants) | 201 | 205
  Change baseline to 3-month follow-up | -0.1 (4.9) | 0.4 (5.3)
  Change baseline to 6-month follow-up: number analyzed (Participants) | 205 | 202
  Change baseline to 6-month follow-up | 0.3 (5.3) | 1.0 (5.0)
  Change baseline to 12-month follow-up: number analyzed (Participants) | 199 | 197
  Change baseline to 12-month follow-up | 0.9 (5.8) | 1.0 (5.3)
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Other; p = 0.21, Mixed Models Analysis; beta coefficient = 0.47, 95% CI 2-sided [-0.27 to 1.22]

10. Secondary Outcome: Reported Services Completed Outside Vanderbilt System
Description: The number of patient reports of diabetes eye exams received outside the Vanderbilt University Medical Center health system submitted via the study intervention.
Time Frame: 12-month follow-up
Population: This analysis is limited to the intervention arm only because only patients in the intervention arm were able to report diabetes eye exams received outside the Vanderbilt University Medical Center health system using the study intervention.
Measure: Number; unit: reports
Arm/Group | Intervention
Number analyzed (Participants) | 216
reports | 101

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 1/217 | 0/216
Serious Adverse Events (participants affected / at risk) | 7/217 | 7/216
Other Adverse Events (participants affected / at risk) | 0/217 | 0/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=217) | Intervention (N=216)
Hospitalization (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 2 (2) | 1 (2)
Hospitalization (Infections and infestations) | 1 (1) | 2 (2)
Hospitalization (Nervous system disorders) | 1 (1) | 2 (5)
Hospitalization (Cardiac disorders) | 2 (6) | 2 (2)
Death (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — motor vehicle accident
Hospitalization (General disorders) | 0 (0) | 1 (1)
Hospitalization (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT04894903/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT04894903/ICF_002.pdf